CLINICAL TRIAL: NCT03464903
Title: ALS Reversals: Genetic Analyses (St.A.R. Protocol 2) RDCRN CReATe Protocol #8007
Brief Title: Study of ALS Reversals 2: Genetic Analyses
Acronym: StAR2
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: CReATe Consortium (funded by NIH/NCATS/NINDS) (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00091570; 8007 (Registry Identifier: Rare Disease Clinical Research Network)
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Amyotrophic Lateral Sclerosis; Progressive Muscular Atrophy
Keywords: amyotrophic lateral sclerosis; progressive muscular atrophy; motor neuron disease; ALS reversals; whole genome sequencing
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Muscular Atrophy, Spinal; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to try to understand why reversals of amyotrophic lateral sclerosis (ALS) and primary muscular atrophy (PMA) take place. The study will enroll patients with ALS or PMA reversals to give saliva samples in order to determine if the ALS or PMA reversal is because of certain changes in the genetic code.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is a devastating motor neuron disease that typically causes rapidly progressive muscle weakness, disability and premature death. In spite of a large number of attempted ALS trials, there are no significant disease-modifying therapies for this condition to-date.

There exists a small group of patients who meet diagnostic criteria for ALS or progressive muscular atrophy (PMA), progress for a period of time, and then significantly improve. Some of these "ALS reversals" even make a complete recovery back to normal neurological function. The investigator has independently verified 34 of these cases so far through review of medical records and peer-reviewed literature. These patients are different in their demographics and disease characteristics as compared to patients with more typically progressive ALS. One possible explanation for these cases is that these patients are genetically different than most patients with ALS and that these differences confer a form of disease "resistance". Study of these selected reversal patients may yield valuable clues to endogenous mechanisms of ALS resistance. The concept of genetic conferred ability to resist a disease is not novel. A group of patients who could unexpectedly "control" HIV due to a mutant allele has led to an improved understanding of HIV pathophysiology and a new treatment

This is a pilot case-control study attempting to discover genetic correlates to ALS reversals. The investigator will collect demographics, disease characteristics, pedigree information and saliva samples from ALS reversals. Whole genome DNA will be extracted and sequenced from these saliva samples. The genomes of ALS reversals will then be compared with whole genome sequencing previously completed from a biorepository of de-identified samples of more typically progressive patients with ALS. The study will not save any saliva samples collected as a part of this new protocol for future research.

ELIGIBILITY:
Inclusion Criteria:

1. Prior participation in Documentation of Known ALS Reversals (Duke IRB Pro00076395)
2. Confirmation of ALS or PMA (primary muscular atrophy) diagnosis through medical record review (previously documented in Documentation of Known ALS Reversals protocol)
3. Sustained, robust improvement on at least one objective ALS outcomes measure (ex. ALSFRS-R, FVC, strength testing, EMG) (previously documented in Documentation of Known ALS Reversals protocol)
4. Able to understand English

Exclusion Criteria:

1. History of cognitive impairment severe enough to preclude informed consent, reported by patient on direct questioning or as suspected by research personnel from Documentation of Known ALS Reversals (Duke IRB Pro00076395) study data
2. Prior participation in the Phenotype Genotype and Biomarkers in ALS and Related Disorders (RDCRN #8001) protocol

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be enrolled by invitation only. Potential participants will have had a previously verified diagnosis of ALS or PMA and a verified sustained and robust reversal of disease.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
genetic comparison | 1 day
  comparison of genes of participants with ALS reversals to genes of more typically progressive patients with ALS

SECONDARY OUTCOMES:
factors associated with genes | 1 day
  further genetic analysis for any interaction of demographics, rate of disease progression, or disease characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Bedlack, MD, PhD, Study Chair — Duke Health
Locations (1):
- Duke ALS Clinic / DUSOM Dept of Neurology / DUHS, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Information obtained from this analysis (genotypic data), as well as information about disease signs and symptoms (phenotypic data), will be entered into one or more scientific repositories maintained by organizations such as the New York Genome Center (NYGC) and the Federal Government. One such repository is the Database of Genotypes and Phenotypes (dbGaP), a data repository at the NIH. All data and information will be submitted via a secure transmission process to a high security network within NIH.
  While the information and data resulting from this study may be presented at scientific meetings or published in a scientific journal, your name or other personal information will not be revealed.

REFERENCES:
- [Background] Ozdinler PH, Silverman RB. Treatment of amyotrophic lateral sclerosis: lessons learned from many failures. ACS Med Chem Lett. 2014 Oct 8;5(11):1179-81. doi: 10.1021/ml500404b. eCollection 2014 Nov 13. PMID 25408825
- [Background] http://www.wsj.com/articles/the-mystery-of-als-patients-who-see-improvement-1465845332
- [Background] ALSUntangled Group. ALSUntangled No. 12: Dean Kraft, Energy Healer. Amyotroph Lateral Scler. 2011 Sep;12(5):389-91. doi: 10.3109/17482968.2011.609309. No abstract available. PMID 21981685
- [Background] Harrison D and Bedlack R (unpublished data).
- [Background] Bedlack RS, Vaughan T, Wicks P, Heywood J, Sinani E, Selsov R, Macklin EA, Schoenfeld D, Cudkowicz M, Sherman A. How common are ALS plateaus and reversals? Neurology. 2016 Mar 1;86(9):808-12. doi: 10.1212/WNL.0000000000002251. Epub 2015 Dec 9. PMID 26658909
- [Background] Samson M, Libert F, Doranz BJ, Rucker J, Liesnard C, Farber CM, Saragosti S, Lapoumeroulie C, Cognaux J, Forceille C, Muyldermans G, Verhofstede C, Burtonboy G, Georges M, Imai T, Rana S, Yi Y, Smyth RJ, Collman RG, Doms RW, Vassart G, Parmentier M. Resistance to HIV-1 infection in caucasian individuals bearing mutant alleles of the CCR-5 chemokine receptor gene. Nature. 1996 Aug 22;382(6593):722-5. doi: 10.1038/382722a0. PMID 8751444
- [Derived] Crayle JI, Rampersaud E, Myers JR, Wuu J, Taylor JP, Wu G, Benatar M, Bedlack RS. Genetic Associations With an Amyotrophic Lateral Sclerosis Reversal Phenotype. Neurology. 2024 Aug 27;103(4):e209696. doi: 10.1212/WNL.0000000000209696. Epub 2024 Jul 30. PMID 39079071
- See also: public website advertising the Study of ALS Reversals Program (St.A.R.) and the Replication of ALS Reversals (R.O.A.R.) Program — http://www.alsreversals.com
- See also: public website with reviews of alternative and off-label treatments with the goal of helping people with ALS make more informed decisions about them — http://www.alsuntangled.com